CLINICAL TRIAL: NCT01575808
Title: The Utility of GP1101 Relative to Surgical Bypass in the Treatment of Femoral / Popliteal Arterial Symptomatic Peripheral Arterial Disease
Brief Title: Multi-center Study for Stent Graft System for Peripheral Artery
Acronym: VJH11-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JPS 16-02 / VJH11-01
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Symptomatic PAD; Stenosis; Occlusion
MeSH Terms: conditions — Peripheral Arterial Disease; Constriction, Pathologic; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GP1101 (Experimental): Prospective data collection: Subjects with occlusive disease of the SFA (Superficial Femoral Artery) implanted with GP1101 covered stent graft
  Interventions: Device: GP1101
- Retrospective Surgical Bypass Outcomes (No Intervention): Retrospective data collection (Apr 2012 - Apr 2014) of 68 surgical procedures (performed after Jan 2002) at six Japanese centers used to treat femoral-popliteal artery symptomatic PAD for purposes of establishing the invasiveness control data for hospital stay duration, avoidance of general anesthesia and avoidance of intra-operative transfusion. Eligibility criteria for inclusion werer established to be consistent with the experimental arm.

INTERVENTIONS:
Device: GP1101 — Endovascular stent graft implantation
  Other Names: Gore VIABAHN Endoprosthesis
  Arms: GP1101

SUMMARY:
The utility of GP1101 will be evaluated relative to that of surgical bypass in the treatment of Femoral/Popliteal Arterial Symptomatic Peripheral Arterial Disease. Efficacy will be measured by comparison to a Surgical Bypass Efficacy Goal, and Invasiveness will be measured by comparison to Surgical Bypass data derived from a retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford 2-5 category
* Subject has read, understood and signed written informed consent which has been reviewed and approved by the Institutional Review Board (IRB).
* At least 20 years of age.
* Ankle-brachial index (ABI) in the study limb in the non-invasive lower extremity arterial studies within 30 days prior to study procedure or at the time of study procedure is less than or equal to 0.9, or toe-brachial index (TBI) is less than or equal to 0.5.
* Male, infertile female, or female of child-bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7 days prior to study procedure.
* Projected life expectancy of greater than 2 years.
* The ability to comply with the study protocol, follow-up requirements and required testing.
* Surgical bypass candidate
* Qualifying lesions by angiography

Exclusion Criteria:

* Untreated flow-limiting aortoiliac disease.
* Any previous stenting or surgery in the target vessel(i.e. femoro-popliteal artery).
* Vascular access/catheterization in the target or contralateral limb within 30 days of study enrollment.
* Planned surgery or intervention within 30 days after study procedure.
* Femoral artery or popliteal artery aneurysm > 1.5 X healthy adjacent vessel diameter.
* Non-atherosclerotic disease resulting in stenosis and/or occlusion (e.g., embolism, Buerger's disease, vasculitis).
* Severe medical comorbidities (untreated CAD/CHF (Congestive Heart Failure), severe COPD (Chronic Obstructive Pulmonary Disease), severe dementia, NYHA (New York Heart Association) 3/4, severe hypertension, etc.)
* Any medical condition that would preclude post-procedural ambulation or completion of study follow-up.
* Rutherford 5 patients with active infection.
* Serum creatinine >2.5 mg/dL within 30 days prior to study procedure.
* Rutherford 6 category in the study or non-study limb or major tissue loss extending above the proximal phalanx level.
* Rutherford 5 characteristics in non-study limb.
* Major distal amputation (above the transmetatarsal) in the study or non-study limb.
* Active infection that could adversely impact patient outcomes in the study, or any patient with septicemia or bacteremia.
* Any previously known coagulation disorder, including hypercoagulability.
* Morbid obesity or operative scarring that precludes percutaneous approach
* Contraindication to anticoagulation or antiplatelet
* Known allergies to stent/stent-graft components, including heparin sensitivity, allergy, or previous incidence of heparin-induced thrombocytopenia (HIT) type II.
* Current peritoneal or hemodialysis
* Participation in another clinical trial (except F/P device clinical trial) up to 3 months prior to study enrollment.
* Enrollment in a F/P device clinical trial within the last 12 months.
* Interventional or surgical treatment on arteries distal to the target vessel for this study within the past 12 months.
* Any other factor identified by the Principal Investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takao Ohki, MD, Principal Investigator — Jikei Medical University Hospital
Locations (15):
- Japan (15):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Shinshu University Hospital, Nagano, Asahi, Matsumoto
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Tokeidai Memorial Hospital, Sapporo, Hokkaido
  - Kansai Rousai Hospital, Amagasaki, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kobe Rosai Hospital, Kobe, Hyōgo
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - National Hospital Organaization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Nara Medical University Hospital, Nara
  - Jikei Medical University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ohki T, Kichikawa K, Yokoi H, Iida O, Yamaoka T, Maeda K, Kanaoka Y. Long-term results of the Japanese multicenter Viabahn trial of heparin bonded endovascular stent grafts for long and complex lesions in the superficial femoral artery. J Vasc Surg. 2021 Dec;74(6):1958-1967.e2. doi: 10.1016/j.jvs.2021.05.056. Epub 2021 Jun 26. PMID 34182032
- [Derived] Ohki T, Kichikawa K, Yokoi H, Uematsu M, Yamaoka T, Maeda K, Kanaoka Y. Outcomes of the Japanese multicenter Viabahn trial of endovascular stent grafting for superficial femoral artery lesions. J Vasc Surg. 2017 Jul;66(1):130-142.e1. doi: 10.1016/j.jvs.2017.01.065. Epub 2017 Apr 8. PMID 28400218

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 133 participants were enrolled into the GP1101 arm; 14 were training cases, 16 were excluded by the Case Conference Committee; total participants started was 103. Retrospective Surgical Bypass Outcomes represent historical controls (n=68).
Groups:
- GP1101: Subjects with occlusive disease of the SFA (Superficial Femoral Artery) implanted with GP1101 covered stent graft >
  > GP1101: Endovascular Device Implantation
- Retrospective Surgical Bypass Outcomes: Retrospective data collection (Apr 2012 - Apr 2014) surgical procedures (performed after Jan 2002) at six Japanese centers used to treat femoral-popliteal artery symptomatic PAD for purposes of establishing the invasiveness control data for hospital stay duration, avoidance of general anesthesia and avoidance of intra-operative transfusion. Eligibility criteria for inclusion were established to be consistent with the experimental arm.
Period: Overall Study
Arm/Group | GP1101 | Retrospective Surgical Bypass Outcomes
Started | 103 | 68
Completed | 100 (Study ongoing. All 103 assessed for primary invasiveness endpoints,100 for primary efficacy endpoint) | 68
Not Completed | 3 | 0
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Retrospective Surgical Bypass Outcomes: Retrospective data collection (Apr 2012 - Apr 2014) of 68 surgical procedures (performed after Jan 2002) at six Japanese centers used to treat femoral-popliteal artery symptomatic PAD for purposes of establishing the invasiveness control data for hospital stay duration, avoidance of general anesthesia and avoidance of intra-operative transfusion. Eligibility criteria for inclusion were established to be consistent with the experimental arm.
- Total: Total of all reporting groups
Arm/Group | GP1101 | Retrospective Surgical Bypass Outcomes | Total
Number analyzed (Participants) | 103 | 68 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (7.0) | 72.3 (8.3) | 73.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 85 | 51 | 136
Region of Enrollment [Number; unit: participants]
  Japan | 103 | 68 | 171
Height [Mean (Standard Deviation); unit: centimeter] — Population: Height was not measured in the Retrospective Surgical Bypass Outcomes arm
  centimeter
    number analyzed (Participants) | 103 | 0 | 103
    (all) | 161.9 (8.48) |  | 161.9 (8.48)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Weight was not measured in the Retrospective Surgical Bypass Outcomes arm
  kilograms
    number analyzed (Participants) | 103 | 0 | 103
    (all) | 59.2 (10.03) |  | 59.2 (10.03)
BMI [Mean (Standard Deviation); unit: kg/㎡] — Body Mass Index Population: BMI was not measured in the Retrospective Surgical Bypass Outcomes arm
  kg/㎡
    number analyzed (Participants) | 103 | 0 | 103
    (all) | 22.5 (2.83) |  | 22.5 (2.83)
Smoking History [Count of Participants; unit: Participants]
  Current Smoker | 29 | 23 | 52
  Not a Current Smoker | 74 | 45 | 119
Diabetes Mellitus [Count of Participants; unit: Participants]
  History of Diabetes Mellitus = Yes | 62 | 34 | 96
  History of Diabetes Mellitus = No | 41 | 34 | 75
Hypertension [Count of Participants; unit: Participants]
  History of Hypertension = Yes | 91 | 59 | 150
  History of Hypertension = No | 12 | 9 | 21
Dyslipidemia [Count of Participants; unit: Participants]
  History of Dyslipidemia = Yes | 64 | 32 | 96
  History of Dyslipidemia = No | 39 | 36 | 75
Carotid Disease [Count of Participants; unit: Participants]
  History of Carotid Disease = Yes | 13 | 6 | 19
  History of Carotid Disease = No | 90 | 62 | 152
Coronary Artery Disease [Count of Participants; unit: Participants]
  History of Coronary Artery Disease = Yes | 42 | 21 | 63
  History of Coronary Artery Disease = No | 61 | 47 | 108
Myocardial Infarction [Count of Participants; unit: Participants]
  History of Myocardial Infarction = Yes | 12 | 7 | 19
  History of Myocardial Infarction - No | 91 | 61 | 152
Congestive Heart Failure [Count of Participants; unit: Participants]
  History of Congestive Heart Failure = Yes | 4 | 3 | 7
  HIstory of Congestive Heart Failure = No | 99 | 65 | 164
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants]
  History of COPD = Yes | 10 | 4 | 14
  History of COPD = No | 93 | 64 | 157
Study Limb [Count of Participants; unit: Participants]
  Right | 56 | 32 | 88
  Left | 47 | 36 | 83
Ankle Brachial Index (ABI) [Mean (Standard Deviation); unit: Ratio] — Population: Eligibility met by TBI for one subject.
  Ratio
    number analyzed (Participants) | 102 | 68 | 170
    (all) | 0.64 (0.12) | 0.47 (0.20) | 0.57 (0.18)
Rutherford Category [Count of Participants; unit: Participants]
  Category 0 - Asymptomatic | 0 | 0 | 0
  Category 1 - Mild Claudication | 0 | 0 | 0
  Category 2 - Moderate Claudication | 45 | 7 | 52
  Category 3 - Severe Claudication | 55 | 44 | 99
  Category 4 - Ischemic Rest Pain | 1 | 7 | 8
  Category 5 - Minor Tissue Loss | 2 | 10 | 12
  Category 6- Major Tissue Loss | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Assisted Patency
Description: Primary Efficacy Endpoint >
  > Primary assisted patency at 12 months, defined as hemodynamic evidence by Angiography or ultrasound of flow through a device that had not required a Target Lesion Revascularization (TLR) to restore blood flow after total occlusion
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- GP1101: Subjects with occlusive disease of the SFA (Superficial Femoral Artery) implanted with GP1101 covered stent graft >
  > GP1101: Endovascular stent graft implantation
Arm/Group | GP1101
Number analyzed (Participants) | 100
Participants | 91
Statistical Analysis 1: Comparison: GP1101; A literature-based Surgical Bypass Efficacy Goal of 65% was compared to the percentage of subjects maintaining primary assisted patency at 12 months. A one-sided z-test using a Type I error of 5% was performed to test the hypotheses that the 12-month primary assisted patency probability of GP1101 is superior to the SBEG of 65%; Test type: Superiority or Other; p < 0.0001, z-test; One-sided z-test; Percentage = 91, 95% CI 1-sided [lower limit 86.3]

2. Primary Outcome: Duration of Stay
Description: Duration (in days) of post-procedure hospital stay
Time Frame: Up to discharge
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | GP1101 | Retrospective Surgical Bypass Outcomes
Number analyzed (Participants) | 103 | 68
Days | 2.0 [2 to 3] | 12.5 [10 to 14]
Statistical Analysis 1: Comparison: GP1101 vs Retrospective Surgical Bypass Outcomes; Hypothesis is that the post-procedure hospital stay duration for GP1101 is superior to the post-procedure hospital stay for the retrospective surgical bypass group; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Rate of Avoidance of General Anesthesia
Description: Percentage of study subjects avoiding general anesthesia
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | GP1101 | Retrospective Surgical Bypass Outcomes
Number analyzed (Participants) | 103 | 68
Participants | 103 | 17
Statistical Analysis 1: Comparison: GP1101 vs Retrospective Surgical Bypass Outcomes; The hypothesis is that the rate of avoidance of general anesthesia for GP1101 is superior to the rate of avoidance of general anesthesis for the retrospective surgical bypass group; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Percentage = 100, 95% CI 2-sided [96.5 to 100] — Confidence interval calculated with binomial exact method

4. Secondary Outcome: Number of Participants Who Did Not Experience Any Critical Events(Death, Target Vessel Revascularization, Major Amputation of the Target Limb)
Description: Composite endpoint of all subjects experiencing death, target vessel revascularization and/or a major amputation of the target limb (above transmetatarsals) within one month of the index procedure.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | GP1101
Number analyzed (Participants) | 103
Participants | 103
Statistical Analysis 1: Comparison: GP1101; Test type: Superiority or Other; Percentage = 100, 95% CI 2-sided [96.5 to 100.0] — Confidence intervals calculated using the binomial exact method

5. Secondary Outcome: Percent of Participants Not Experiencing an Adverse Event
Description: % Avoidance of serious adverse events that are device or procedure-related or for which the relationship is unknown
Time Frame: 1 month
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- GP1101: Prospective data collection: Subjects with occlusive disease of the SFA (Superficial Femoral Artery) implanted with GP1101 covered stent graft >
  > GP1101: Endovascular stent graft implantation
Arm/Group | GP1101
Number analyzed (Participants) | 103
percent of participants | 97.1 [91.2 to 99.1]

6. Secondary Outcome: Percent of Participants Not Experiencing an Adverse Event
Description: % Avoidance of serious adverse events that are device or procedure-related or for which the relationship is unknown at 12 months.
Time Frame: 3 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | GP1101
Number analyzed (Participants) | 103
Percent of participants | 97.1 [91.2 to 99.1]

7. Secondary Outcome: Percent of Participants Not Experiencing an Adverse Event
Description: % Avoidance of serious adverse events that are device or procedure-related or for which the relationship is unknown
Time Frame: 6 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | GP1101
Number analyzed (Participants) | 103
percent of participants | 95.1 [88.7 to 97.9]

8. Secondary Outcome: Percent of Participants Not Experiencing an Adverse Event
Description: % Avoidance of serious adverse events that are device or procedure-related or for which the relationship is unknown
Time Frame: 12 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | GP1101
Number analyzed (Participants) | 103
percent of participants | 90.9 [82.3 to 95.4]

9. Secondary Outcome: Percent of Participants Not Experiencing an Adverse Event
Description: % Avoidance of serious adverse events that are device or procedure-related or for which the relationship is unknown
Time Frame: 24 months
Reporting Status: Not Posted

10. Secondary Outcome: Percent of Participants Not Experiencing an Adverse Event
Description: % Avoidance of serious adverse events that are device or procedure-related or for which the relationship is unknown
Time Frame: 36 months
Reporting Status: Not Posted

11. Secondary Outcome: Percent of Participants Not Experiencing an Adverse Event
Description: % Avoidance of serious adverse events that are device or procedure-related or for which the relationship is unknown
Time Frame: 48 months
Reporting Status: Not Posted

12. Secondary Outcome: Rate of Avoidance of Adverse Events
Description: % Avoidance of serious adverse events that are device or procedure-related or for which the relationship is unknown
Time Frame: 60 months
Reporting Status: Not Posted

13. Secondary Outcome: Technical Success
Description: Placement of GP1101 with residual stenosis of less than 30%
Time Frame: Post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- GP1101: Prospective data collection: Subjects with occlusive disease of the SFA (Superficial Femoral Artery) implanted with GP1101 covered stent graft>
  > GP1101: Endovascular stent graft implantation
Arm/Group | GP1101
Number analyzed (Participants) | 103
Participants | 102

14. Secondary Outcome: Primary Patency
Description: Hemodynamic blood flow through GP1101 that had not required a target lesion revascularization
Time Frame: 1 month
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 99.0 [93.2 to 99.9]

15. Secondary Outcome: Primary Patency
Description: Hemodynamic blood flow through GP1101 that had not required a target lesion revascularization
Time Frame: 3 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 97.1 [91.2 to 99.0]

16. Secondary Outcome: Primary Patency
Description: Hemodynamic blood flow through GP1101 that had not required a target lesion revascularization
Time Frame: 6 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 92.1 [84.8 to 96.0]

17. Secondary Outcome: Primary Patency
Description: Hemodynamic blood flow through GP1101 that had not required a target lesion revascularization
Time Frame: 12 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 92.1 [84.8 to 96.0]

18. Secondary Outcome: Primary Patency
Description: Hemodynamic blood flow through GP1101 that had not required a target lesion revascularization
Time Frame: 24 months
Reporting Status: Not Posted

19. Secondary Outcome: Secondary Patency
Description: No bypass surgery and no occlusion at the target site
Time Frame: 1 month
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 99.0 [93.2 to 99.9]

20. Secondary Outcome: Secondary Patency
Description: No bypass surgery and no occlusion at the target site
Time Frame: 3 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 98.0 [92.4 to 99.5]

21. Secondary Outcome: Secondary Patency
Description: No bypass surgery and no occlusion at the target site
Time Frame: 6 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 98.0 [92.4 to 99.5]

22. Secondary Outcome: Secondary Patency
Description: No bypass surgery and no occlusion at the target site
Time Frame: 12 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 98.0 [92.4 to 99.5]

23. Secondary Outcome: Secondary Patency
Description: No bypass surgery and no occlusion at the target site
Time Frame: 24 months
Reporting Status: Not Posted

24. Secondary Outcome: Rate of Avoidance of Stent Fracture
Description: X-ray for stent fracture evaluated by Core Lab
Time Frame: 1 month
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 100.0 [100.0 to 100.0]

25. Secondary Outcome: Rate of Avoidance of Stent Fracture
Description: X-ray for stent fracture evaluated by Core Lab
Time Frame: 3 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 100.0 [100.0 to 100.0]

26. Secondary Outcome: Rate of Avoidance of Stent Fracture
Description: X-ray for stent fracture evaluated by Core Lab
Time Frame: 6 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 100.0 [100.0 to 100.0]

27. Secondary Outcome: Rate of Avoidance of Stent Fracture
Description: X-ray for stent fracture evaluated by Core Lab
Time Frame: 12 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 100.0 [100.0 to 100.0]

28. Secondary Outcome: Rate of Avoidance of Stent Fracture
Description: X-ray for stent fracture evaluated by Core Lab
Time Frame: 24 months
Reporting Status: Not Posted

29. Secondary Outcome: Avoidance of Target Lesion Revascularization
Time Frame: 1 month
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 100.0 [100.0 to 100.0]

30. Secondary Outcome: Avoidance of Target Lesion Revascularization
Time Frame: 3 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 99.0 [93.2 to 99.9]

31. Secondary Outcome: Avoidance of Target Lesion Revascularization
Time Frame: 6 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 95.1 [88.6 to 97.9]

32. Secondary Outcome: Avoidance of Target Lesion Revascularization
Time Frame: 12 months
Population: Kaplan-Meier estimate done at end of follow-up visit window
Measure: Number (95% Confidence Interval); unit: Probability of having an event
Arm/Group | GP1101
Number analyzed (Participants) | 103
Probability of having an event | 93.1 [86.1 to 96.7]

33. Secondary Outcome: Avoidance of Target Lesion Revascularization
Time Frame: 24 months
Reporting Status: Not Posted

34. Secondary Outcome: Clinical Success
Description: The Rutherford Classification is a system used to score Chronic Limb Ischemia in Peripheral Artery Disease (PAD). The stages follow (higher numbers are worse):
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
  The percentage of people improving by at least one stage (moving frm higher number to lower number) is listed in the results.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | GP1101
Number analyzed (Participants) | 103
Participants | 100
Statistical Analysis 1: Comparison: GP1101; Test type: Other; Percentage = 97.1, 95% CI 2-sided [91.7 to 99.4]

35. Secondary Outcome: Clinical Success
Description: as for outcome 34
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | GP1101
Number analyzed (Participants) | 102
Participants | 98

36. Secondary Outcome: Clinical Success
Description: as for outcome 34
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | GP1101
Number analyzed (Participants) | 102
Participants | 97

37. Secondary Outcome: Clinical Success
Description: as for outcome 34
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | GP1101
Number analyzed (Participants) | 99
Participants | 90

38. Secondary Outcome: Clinical Success
Description: as for outcome 34
Time Frame: 24 months
Reporting Status: Not Posted

39. Secondary Outcome: Change in Ankle-Brachial Index From Baseline
Description: Ankle-Brachial Index of each time frame (1, 3, 6, 12, 24 months) compared to baseline (pre-procedure),
Time Frame: Baseline and 1, 3, 6, 12, 24 months, change from baseline at 1 month presented
Measure: Mean (Standard Deviation); unit: ABI
Arm/Group | GP1101
Number analyzed (Participants) | 103
ABI | 0.98 (0.118)

40. Secondary Outcome: Change in Ankle-Brachial Index From Baseline
Description: Ankle-Brachial Index of each time frame (1, 3, 6, 12, 24 months) compared to baseline (pre-procedure)
Time Frame: Baseline and 1, 3, 6, 12, 24 months, change from baseline at 3 months presented
Measure: Mean (Standard Deviation); unit: ABI
Arm/Group | GP1101
Number analyzed (Participants) | 101
ABI | 0.97 (0.137)

41. Secondary Outcome: Change in Ankle-Brachial Index From Baseline
Description: Ankle-Brachial Index of each time frame (1, 3, 6, 12, 24 months) compared to baseline (pre-procedure)
Time Frame: Baseline and 1, 3, 6, 12, 24 months, change from baseline at 6 months presented
Measure: Mean (Standard Deviation); unit: ABI
Arm/Group | GP1101
Number analyzed (Participants) | 102
ABI | 0.95 (0.137)

42. Secondary Outcome: Change in Ankle-Brachial Index From Baseline
Description: Ankle-Brachial Index of each time frame (1, 3, 6, 12, 24 months) compared to baseline (pre-procedure)
Time Frame: Baseline and 1, 3, 6, 12, 24 months, change from baseline at 12 months presented
Measure: Mean (Standard Deviation); unit: ABI
Arm/Group | GP1101
Number analyzed (Participants) | 94
ABI | 0.94 (0.171)

43. Secondary Outcome: Change in Ankle-Brachial Index From Baseline
Description: Ankle-Brachial Index of each time frame (1, 3, 6, 12, 24 months) compared to baseline (pre-procedure)
Time Frame: Baseline and 1, 3, 6, 12, 24 months, change from baseline at 24 months presented
Reporting Status: Not Posted

44. Secondary Outcome: Vascular Quality of Life Questionnaire - VascuQOL
Description: VascuQOL Score - Higher score reflects a better quality of life(Score range: 1 to 7). This score is composed of "Activity", "Symptom", "Pain", "Emotional" and "Social" scores as subscales. The total score is calculated as the average value of all scores.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GP1101
Number analyzed (Participants) | 103
units on a scale | 5.5 (1.09)

45. Secondary Outcome: Vascular Quality of Life Questionnaire - VascuQOL
Description: as for outcome 44
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GP1101
Number analyzed (Participants) | 101
units on a scale | 5.3 (1.26)

46. Secondary Outcome: Vascular Quality of Life Questionnaire - VascuQOL
Description: as for outcome 44
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GP1101
Number analyzed (Participants) | 102
units on a scale | 5.3 (1.23)

47. Secondary Outcome: Vascular Quality of Life Questionnaire - VascuQOL
Description: as for outcome 44
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GP1101
Number analyzed (Participants) | 94
units on a scale | 5.1 (1.30)

48. Secondary Outcome: Vascular Quality of Life Questionnaire - VascuQOL
Description: as for outcome 44
Time Frame: 24 months
Reporting Status: Not Posted

49. Secondary Outcome: Walking Impairment Questionnaire-WIQ
Description: WIQ Distance Score - Higher score reflects a better quality of life（Scores range: 0 to 100.）The difficulty of walking with each specific distance(from walking indoor to 450 meter) is ranked on 0 to 4 and these rank value are converted to score according to the difficulty of walking. The distance score is determained by dividing the total score by greatest score and multiplying by 100.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GP1101
Number analyzed (Participants) | 103
units on a scale | 66.9 (34.2)

50. Secondary Outcome: Walking Impairment Questionnaire-WIQ
Description: as for outcome 49
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GP1101
Number analyzed (Participants) | 101
units on a scale | 63.9 (34.0)

51. Secondary Outcome: Walking Impairment Questionnaire-WIQ
Description: as for outcome 49
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GP1101
Number analyzed (Participants) | 102
units on a scale | 67.0 (34.1)

52. Secondary Outcome: Walking Impairment Questionnaire-WIQ
Description: as for outcome 49
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GP1101
Number analyzed (Participants) | 94
units on a scale | 64.0 (34.5)

53. Secondary Outcome: Walking Impairment Questionnaire-WIQ
Description: as for outcome 49
Time Frame: 24 months
Reporting Status: Not Posted

54. Secondary Outcome: Rate of Avoidance of Blood Transfusion
Time Frame: Post-Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | GP1101
Number analyzed (Participants) | 103
Participants | 103
Statistical Analysis 1: Comparison: GP1101; Test type: Other; Percentage = 100, 95% CI 2-sided [96.5 to 100.0] — Confidence Interval calculated with binomial exact method

ADVERSE EVENTS:
Description: Adverse events were systematically reported on Case Report Forms
Arm/Group | GP1101
Serious Adverse Events (participants affected / at risk) | 47/103
Other Adverse Events (participants affected / at risk) | 41/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GP1101 (N=103)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Angina pectoris aggravated (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Anginal attack (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrial fibrillation paroxysmal (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 3
Non-sustained ventricular tachycardia (Cardiac disorders) | 1
Bilateral cataracts (Eye disorders) | 1
Cataract aggravated (Eye disorders) | 1
Left cataract (Eye disorders) | 1
Right cataract (Eye disorders) | 1
Acute gastritis (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Haemorrhage of digestive tract (Gastrointestinal disorders) | 1
Right inguinal hernia (Gastrointestinal disorders) | 1
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1
Adverse drug reaction (General disorders) | 1
Arterial stent occlusion (General disorders) | 2
Chest pain (General disorders) | 1
Device occlusion (General disorders) | 7
Hepatic function disorder (Hepatobiliary disorders) | 1
Allergic reaction to antibiotics (Immune system disorders) | 1
Acute pneumonia (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza A virus infection (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pulmonary aspergillosis (Infections and infestations) | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 1
Chronic subdural haematoma (Injury, poisoning and procedural complications) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1
In-stent peripheral artery restenosis (Injury, poisoning and procedural complications) | 10
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Malleolar fracture (Injury, poisoning and procedural complications) | 1
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1
Poisoning by hypnotic (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
CRP increased (Investigations) | 1
Potassium abnormal (Investigations) | 1
Sugar blood level increased (Investigations) | 1
Insulin hypoglycaemia (Metabolism and nutrition disorders) | 1
Loss of control of blood sugar (Metabolism and nutrition disorders) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant neoplasm of lateral wall of oropharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope vasovagal (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Renal failure chronic aggravated (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Femoral artery occlusion (Vascular disorders) | 1
Iliac artery stenosis (Vascular disorders) | 4
Peripheral artery stenosis (Vascular disorders) | 1
Thromboembolism (Vascular disorders) | 1
Vascular occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GP1101 (N=103)
Adverse drug reaction (General disorders) | 10
Implant site pain (General disorders) | 18
Pyrexia (General disorders) | 8
Vessel puncture site pain (General disorders) | 6
Common cold (Infections and infestations) | 6
Hypertension aggravated (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No